CLINICAL TRIAL: NCT07301671
Title: Prospective Longitudinal Observational Cohort Study of a Digital Automated Rehabilitation Model for Shoulder Disorders (REHABI) in a Private Physiotherapy Clinic
Brief Title: Prospective Cohort of Digital Shoulder Rehabilitation Using the REHABI System in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: Universidad Pública de Navarra (Other)
Collaborators: Gobierno de Navarra (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1479272TES; 0011-1408-2022-000012 (Other: Beca de Doctorado Industrial 2022 del Gobierno de Navarra)
Record Dates: First submitted 2025-11-26; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Digital Shoulder Rehabilitation
Keywords: Shoulder rehabilitation; digital physiotherapy; functional assessment; responsiveness (SRM); clinical effectiveness; Clinical automation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective longitudinal observational cohort study of patients with shoulder disorders undergoing a standardized rehabilitation program supported by the REHABI digital automated model in a private physiotherapy clinic. The study aims to describe clinical outcomes in routine practice and to optimize a 24-test functional assessment battery based on deficit prevalence, magnitude, and responsiveness.

DETAILED DESCRIPTION:
This is a prospective longitudinal observational cohort study of 129 adult patients (≥18 and ≤71 years) with acute non-traumatic shoulder pain and/or dysfunction treated in a private sports physiotherapy clinic in Pamplona, Spain. All patients undergo a standardized rehabilitation program supported by the REHABI automated digital model, which links quantified deficits obtained from a 24-test functional assessment battery to specific exercise prescriptions and progression rules. The study aims to describe clinical outcomes in routine practice (global clinical deficit score, shoulder pain intensity, number of treatment sessions, and days to discharge) and to optimize the initial 24-test battery based on deficit prevalence, magnitude, and responsiveness to change between baseline and discharge.

The main objectives are: (1) to evaluate the clinical effectiveness and feasibility of the REHABI model in routine clinical practice; and (2) to reduce the initial 24-test assessment battery to a smaller core set of tests using mixed criteria based on prevalence, magnitude of deficit, and responsiveness to change.

ELIGIBILITY:
Inclusion Criteria:

* 18-71 years of age, acute non-traumatic shoulder pain/dysfunction, and access to a smartphone to view the exercises.

Exclusion Criteria:

* Acute fractures or dislocations, arthritis/arthrosis, osteosarcoma, osteomyelitis, and recent shoulder surgeries.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with musculoskeletal shoulder pain treated in a private sports physiotherapy clinic in Pamplona, Spain, who are referred or self-referred for conservative management, consecutively enrolled in the REHABI digital rehabilitation program, and who have access to and basic skills to use a smartphone.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Change in global clinical deficit score from baseline to discharge | Baseline and discharge (approximately 1-6 months after baseline, depending on clinical evolution)
  Global clinical score summarizing the number and magnitude of positive findings in the functional test battery. Higher scores indicate greater functional deficit. Change is calculated as discharge score minus baseline score.

SECONDARY OUTCOMES:
Change in selected functional tests from the optimized core battery | Baseline and discharge (ranging from 1 month to 6 month after baseline)
  Change in performance on selected shoulder functional tests (e.g., Yocum, Speed, Jobe, external rotation at 90° abduction, etc.) identified as part of the optimized core test battery.
Number of rehabilitation sessions until discharge | From baseline to discharge (approximately 1-6 months)
  Total number of physiotherapy sessions attended from baseline to discharge within the REHABI program.
Days from baseline to clinical discharge | Baseline to discharge (ranging from 1 to 6 months)
  Number of days between the first assessment and the discharge visit recorded in the REHABI system.
Change in shoulder pain intensity (Numeric Rating Scale, 0-10) | Baseline and discharge (approximately 1-6 months)
  Shoulder pain intensity during movement, measured using an 11-point Numeric Rating Scale (EVA 0-10). Change is calculated as discharge score minus baseline score.

CONTACTS AND LOCATIONS:
Overall Officials: Lorena Y Castaño, PhD student, Principal Investigator — Universidad Publica de Navarra; Igor Setuain, Phd, Study Director — TDN Clinica; Jose A Sanz D, PhD, Study Director — Universidad Publica de Navarra; Iban Latasa Z., PhD, Study Director — IED Electronics
Locations (1):
- Lorena Castaño de Egues, Noáin, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No
At present, there is no plan to share individual participant data (IPD). This is a single-center study with a relatively small sample and detailed clinical assessments, which may increase the risk of re-identification, and the original informed consent did not explicitly cover broad IPD sharing. De-identified summary results will be available in the published manuscript, and additional aggregated information may be considered upon reasonable request.

REFERENCES:
- [Result] Setuain I, Gonzalez-Izal M, Paularena A, Luque JL, Andersen LL, Izquierdo M. A protocol for a new methodological model for work-related shoulder complex injuries: From diagnosis to rehabilitation. BMC Musculoskelet Disord. 2017 Feb 7;18(1):70. doi: 10.1186/s12891-017-1435-2. PMID 28173784